CLINICAL TRIAL: NCT05716022
Title: Hiatal Hernia and Pulmonary Involvement Related to Subclinical Lung Injury and Fibrosis
Brief Title: Hiatal Hernia and Pulmonary Involvement
Status: Active, not recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: American College of Chest Physicians (Other)
Responsible Party: Principal Investigator, John Kim, MD, MS, Assistant Professor, University of Virginia
Other Study IDs: HSR220294
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Hiatal Hernia; Interstitial Lung Disease
Keywords: Hiatal Hernia; BALF; Interstitial lung Disease
MeSH Terms: conditions — Hernia, Hiatal; Lung Diseases, Interstitial | interventions — Blood Specimen Collection; Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid samples Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hiatal Hernia Group: The subject has a history of acid reflux and/or hiatal hernia undergoing surgical repair by thoracic surgery at the University of Virginia.
  Interventions: Diagnostic Test: Blood Collection; Diagnostic Test: Bronchoscopy
- Control Group: Patients undergoing bronchoscopy for clinical purposes at the University of Virginia endoscopy suite without a clinical diagnosis of hiatal hernia and/or pulmonary fibrosis.
  Interventions: Diagnostic Test: Blood Collection; Diagnostic Test: Bronchoscopy

INTERVENTIONS:
Diagnostic Test: Blood Collection — Prior to subject's surgical procedure, blood (about 3 tablespoons (44 mL)) will be collected through a needle in vein for research purposes. The UVA researchers will analyze the biomarkers that are expressed in subject's blood.
Diagnostic Test: Bronchoscopy — Following blood collection, the subject will undergo the bronchoscopy for research purposes. While in the operating room, a bronchoscope will be inserted through the breathing tube that is already been placed for the surgery. Subject's airways will be examined with the bronchoscope in both lungs. Ten tablespoons (150 mL) of saline solution will be injected into one of subject airways. The fluid will be re-collected by suctioning it back up with the bronchoscope. The fluid will be collected from the bronchscope.

SUMMARY:
Patients often present with a significant burden of fibrosis upon diagnosis as there is interest in identifying these individuals earlier in their disease course (i.e., "subclinical disease") where targeted treatments and modification of risk factors may curb their progression to fulminant fibrosing ILD. The investigators have investigated with computed tomography (CT) methods such as interstitial lung abnormalities (ILA) and high attenuation areas (HAAs) that may detect early radiological signs of interstitial lung inflammation and scarring and novel modifiable risk factors that contribute to its pathogenesis. Among adults without clinically-diagnosed pulmonary fibrosis, those with a hiatal hernia will have higher levels of pepsin in bronchoalveolar lavage fluid (BALF) compared with adults without a hiatal hernia. Secondarily, examinination on whether there are differences in other reflux contents from BALF including total bile, and peripheral biomarkers related to lung injury and fibrogenesis which include matrix metalloproteinase-7 (MMP-7), vascular cell adhesion molecule 1 (VCAM-1), and cancer antigen 125 (CA-125).

DETAILED DESCRIPTION:
Fibrosing interstitial lung diseases (ILDs) have significant morbidity and poor overall survival as the investigation of earlier stages of fibrosing ILDs may identify modifiable risk factors and elucidate its pathogenesis. Interstitial lung disease (ILD) constitutes a group of chronic respiratory illnesses that are characterized by repetitive injury to the lung parenchyma that may progress to fibrosis. Fibrosing ILDs, which include idiopathic pulmonary fibrosis (IPF) and other ILD types, can lead to chronic respiratory failure, and poor survival, is the most common indication for lung transplantation. While antifibrotics slow disease progression and may reduce mortality, they carry side effects and are frequently poorly tolerated by patients. Therefore, there is a critical need to identify novel therapeutic targets. Patients often present with a significant burden of fibrosis upon diagnosis as there is interest in identifying these individuals earlier in their disease course (i.e., "subclinical disease") where targeted treatments and modification of risk factors may curb their progression to fulminant fibrosing ILD.

Hiatal hernia and its promotion of gastroesophageal reflux have been implicated as a causal risk factor in pulmonary fibrosis. One potential modifiable risk factor is hiatal hernia and its promotion of gastroesophageal reflux (GER). Gastric materials in the lung induce parenchymal injury and fibrosis in pre-clinical models as GER may be a vehicle of repetitive lung injury that is then followed by aberrant wound healing and eventual fibrosis. Hiatal hernia, which is the protrusion of stomach contents in the thoracic cavity, can promote GER and is more prevalent in adults with pulmonary fibrosis compared with healthy controls and other chronic lung diseases. Further evidence comes from studies in which patients with IPF and other fibrosing ILDs (many of whom had a hiatal hernia) demonstrated elevated levels of pepsin in their bronchoalveolar lavage fluid (BALF), a significant component of reflux and measurable biomarker, compared with healthy controls and is associated with a higher risk of exacerbation. Much of these studies have been case-control and performed in adults with clinically-diagnosed fibrosing ILD which limits causal inferences. It has been hypothesized that fibrosis itself may promote GER due to impaired esophageal sphincter function due to reduced elasticity and more negative intrathoracic pressures. Whether hiatal hernia contributes to subclinical repetitive injury to the lung among adults without clinically-diagnosed ILD is a significant knowledge gap.

Overactivation of the mononuclear phagocyte immune system may contribute to developing fibrosing ILDs and their progression. Single-cell RNA sequencing (scRNA-seq) has accelerated our understanding of fibrosing ILD by identifying biological pathways related to certain cellular populations. Using scRNA-seq, our group and others have demonstrated that overactivation of the mononuclear phagocyte system, a key component of the innate immune system, may be critical in the pathogenesis of IPF with higher populations of monocytes found in the lungs and blood of patients with fibrosis. Higher levels of the absolute monocyte count in the blood are associated with disease progression and worse survival among adults with IPF. The investigators have extended these findings to earlier stages of ILD as higher monocyte counts are associated with more ILA and its progression on CT and a lower forced vital capacity. Notably, adults with ILA have more activated monocytes than those without ILA, suggesting a smoldering activation of innate immunity may prime an individual to developing ILD in combination with other risk factors (i.e., smoking, genetic variants, and hiatal hernia).

Radiologically-detected hiatal hernia is associated with a greater burden of CT interstitial lung abnormalities and worse survival among community-dwelling adults. In a population cohort of U.S. community-dwelling adults, investigators found that the presence of hiatal hernia on CT was associated with more HAAs and their progression over time and more ILA among younger adults. Notably, elevated HAAs on CT were associated with worse survival among those with a hiatal hernia compared with those without a hernia. Our findings suggest that hiatal hernia and its promotion of GER may contribute to subclinical injury and remodeling detected by imaging biomarkers. Whether subclinical abnormalities are detected in the lungs of adults with hiatal hernia remains a major knowledge gap that this study will address by examining BALF contents of adults with hiatal hernia.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written consent.
2. Clinical diagnosis of hiatal hernia and/or gastroesophageal reflux undergoing pre-operative evaluation for surgical repair at the University of Virginia as part of clinical care.
3. 18 years and above.

Exclusion Criteria:

1. Unable to provide written consent.
2. Clinical diagnosis of pulmonary fibrosis.
3. History of hiatal hernia (for control group only).
4. Use of home supplemental oxygen therapy either at rest or exertion.
5. Pregnant Women (will be confirmed as part of standard of care).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Participants without a clinical diagnosis of pulmonary fibrosis will be recruited from UVA medical center based on the absence of traction bronchiectasis, honeycombing and/or reticular opacities on CT Scan.
  2. Case group will be adults who have a clinical diagnosis of hiatal hernia already scheduled to under surgical repair
  3. Control group will be adults without a CT diagnosis of hiatal hernia who have been scheduled to undergo Bronchoscopy for lung nodule evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bronchoalveolar lavage fluid pepsin levels | Baseline
  Investigators examine whether bronchoalveolar lavage fluid levels of pepsin are significantly different by case (adults with hiatal hernia and/or gastroesophageal reflux undergoing surgical repair) and control status (adults without hiatal hernia). Pepsin levels will be measured by ELISA assay.

SECONDARY OUTCOMES:
Serum matrix metalloproteinase-7 | Baseline
  Serum matrix metalloproteinase-7 will be measured by ELISA assay.
Serum CA-125 | Baseline
  Serum CA-125 will be measured by ELISA assay.
Serum vascular cell adhesion molecule-1 | Baseline
  Serum vascular cell adhesion molecule-1 will be measured by ELISA assay.
RNA gene expression | Baseline
  Gene set enrichment analysis (GSEA) will be performed with a false-discovery rate of <5%. GSEA uses a priori sets of genes that have been grouped together by their common biological pathway stored in databases. Genes constituting very high and low expression will be determined by using the R package "GOSim" with a cutoff q-value <0.01. Cell Population Mapping will be used, an algorithm in the R package "scBio", to perform cell composition analysis and determine the relative abundance of cell compositions. Reference RNA-seq dataset from healthy donors with an annotated cell type meta data from the Broad Institute Single Cell Portal will be used.

CONTACTS AND LOCATIONS:
Overall Officials: John Kim, MD, Principal Investigator — University of Virginia; Roselove Asare, MA, Study Director — UVA; Yousef Althulth, MD, Study Director — UVA
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will become available 24 months after completion of study upon request to principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Will become available 24 months after completion of study upon request to principal investigator.

REFERENCES:
- [Background] Kim JS, Kim J, Yin X, Hiura GT, Anderson MR, Hoffman EA, Raghu G, Noth I, Manichaikul A, Rich SS, Smith BM, Podolanczuk AJ, Garcia CK, Barr RG, Prince MR, Oelsner EC. Associations of hiatus hernia with CT-based interstitial lung changes: the MESA Lung Study. Eur Respir J. 2023 Jan 27;61(1):2103173. doi: 10.1183/13993003.03173-2021. Print 2023 Jan. PMID 35777776
- [Background] Kim JS, Axelsson GT, Moll M, Anderson MR, Bernstein EJ, Putman RK, Hida T, Hatabu H, Hoffman EA, Raghu G, Kawut SM, Doyle MF, Tracy R, Launer LJ, Manichaikul A, Rich SS, Lederer DJ, Gudnason V, Hobbs BD, Cho MH, Hunninghake GM, Garcia CK, Gudmundsson G, Barr RG, Podolanczuk AJ. Associations of Monocyte Count and Other Immune Cell Types with Interstitial Lung Abnormalities. Am J Respir Crit Care Med. 2022 Apr 1;205(7):795-805. doi: 10.1164/rccm.202108-1967OC. PMID 34929108
- [Background] Scott MKD, Quinn K, Li Q, Carroll R, Warsinske H, Vallania F, Chen S, Carns MA, Aren K, Sun J, Koloms K, Lee J, Baral J, Kropski J, Zhao H, Herzog E, Martinez FJ, Moore BB, Hinchcliff M, Denny J, Kaminski N, Herazo-Maya JD, Shah NH, Khatri P. Increased monocyte count as a cellular biomarker for poor outcomes in fibrotic diseases: a retrospective, multicentre cohort study. Lancet Respir Med. 2019 Jun;7(6):497-508. doi: 10.1016/S2213-2600(18)30508-3. Epub 2019 Mar 29. PMID 30935881
- [Background] Wijsenbeek M, Cottin V. Spectrum of Fibrotic Lung Diseases. N Engl J Med. 2020 Sep 3;383(10):958-968. doi: 10.1056/NEJMra2005230. No abstract available. PMID 32877584
- [Background] Lee JS, Song JW, Wolters PJ, Elicker BM, King TE Jr, Kim DS, Collard HR. Bronchoalveolar lavage pepsin in acute exacerbation of idiopathic pulmonary fibrosis. Eur Respir J. 2012 Feb;39(2):352-8. doi: 10.1183/09031936.00050911. Epub 2011 Dec 19. PMID 22183478
- [Background] Noth I, Zangan SM, Soares RV, Forsythe A, Demchuk C, Takahashi SM, Patel SB, Strek ME, Krishnan JA, Patti MG, Macmahon H. Prevalence of hiatal hernia by blinded multidetector CT in patients with idiopathic pulmonary fibrosis. Eur Respir J. 2012 Feb;39(2):344-51. doi: 10.1183/09031936.00099910. Epub 2011 Jul 7. PMID 21737563